CLINICAL TRIAL: NCT02947815
Title: A Randomized, Double Blind, Multi-center, Active Drug Controlled, Phase II/III Clinical Trial to Compare the Safety and Efficacy of NABOTA Versus BOTOX in Treatment of Essential Blepharospasm
Brief Title: Safety and Efficacy of NABOTA in Treatment of Essential Blepharospasm
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWP450007
Record Dates: First submitted 2016-10-24; First posted 2016-10-28 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Blepharospasm
MeSH Terms: conditions — Blepharospasm | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NABOTA (Experimental): Single-dose
  Interventions: Drug: Clostridium Botulinum Toxin Type A
- BOTOX (Active Comparator): Single-dose
  Interventions: Drug: Clostridium Botulinum Toxin Type A

INTERVENTIONS:
Drug: Clostridium Botulinum Toxin Type A
  Other Names: NABOTA
  Arms: NABOTA
Drug: Clostridium Botulinum Toxin Type A
  Other Names: BOTOX
  Arms: BOTOX

SUMMARY:
The purpose of this study is to evaluate the Efficacy and Safety of NABOTA in treatment of essential blepharospasm

ELIGIBILITY:
Inclusion Criteria:

* Male of female of at least 18 years old
* Grade 2~4 in Scott's scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
The change from baseline in Scott's Scale Score | At 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- the catholic university of korea, Seoul ST. Mary's Hospital., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No